## Title:

Study Protocol and Statistical Analysis Plan
The Effect of Simple Basal Insulin Titration,
Metformin Plus Liraglutide for Type 2
Diabetes With Very Elevated HbA1c - The
SIMPLE Study

## **NCT Number:**

NCT01966978

**Date of the Document:** 

05/06/2017

| 1 | |
|---|---|
| 2 | SIMPLE STUDY: SIMPLE BASAL INSULIN |
| 3 | TITRATION, METFORMIN PLUS |
| 4 | LIRAGLUTIDE FOR TYPE 2 DIABETES WITH |
| 5 | VERY ELEVATED HBA1C |
| 6 | |
| 7 | (A RANDOMIZED TRIAL COMPARING THE EFFICACY, SAFETY, AND |
| 8 | HEALTHCARE RELATED COSTS OF TREATING PATIENTS WITH VERY |
| 9 | ELEVATED HBA1c LEVELS WITH BASAL-BOLUS INSULIN REGIMEN OR BASAL |
| 10 | INSULIN WITH A GLP-1 AGONIST) |
| 11 | INSOLIN WITH A GLI -1 MOONIST) |
| 12 | |
| 13 | |
| 14 | INVESTIGATOR-INITIATED STUDY PROPOSAL |
| 15 | FUNDING PROVIDED BY NOVONORDISK A/S |
| 16 | |
| 17 | |
| 18 | UNIVERSAL TRIAL NUMBER (UTN) |
| 19 | U1111-1145-7585 |
| 20 | |
| 21 | |
| 22<br>23 | |
| 24 | |
| 25 | Department of Internal Medicine – Division of Endocrinology and Diabetes |
| 26 | UT Southwestern Medical Center |
| 27 | 5323 Harry Hines Blvd. Dallas, TX 75390-8857 |
| 28 | |
| 29 | |
| 30 | Correspondence to: |
| 31 | Ildiko Lingvay, MD, MPH, MSCS |
| 32 | Associate Professor |
| 33 | UT Southwestern Medical Center, Division of Endocrinology |
| 34 | 5323 Harry Hines Blvd 75390-8857 |
| 35<br>36 | 214-648-2779 |
| 36<br>37 | Ildiko.Lingvay@UTSouthwestern.edu |
| 51 | |

#### **BACKGROUND AND SIGNIFICANCE:**

40 <u>1. Achieving glycemic goals in type 2 diabetes has multiple beneficial health</u>
 41 <u>consequences.</u>

There are over 25 million patients with diabetes in the US [1], a disease with tremendous health, social, and economic implications. Studies like UKPDS [2, 3] and Kumamoto [4, 5] have established an undeniable link between hyperglycemia and micro- and even macrovascular complications. Such data serves as the background for the current glycemic targets recommended by the American Diabetes Association. Despite tremendous therapeutic advances and availability of numerous new classes of drugs in the past decade, more than a third of the population with diabetes, particularly in minority groups and those with lower level of education, still does not reach glycemic targets [6-8]. Given the large epidemic of obesity and type 2 diabetes, our efforts to curb diabetes related morbidity and mortality have a whole new meaning and huge potential impact, both on patient related outcomes as well as cost of healthcare – a very timely concern for our healthcare system[9-11].

## 2. Treatment guidelines for type 2 diabetes advocate insulin treatment for patients with a HbA1c>10%.

Treatment guidelines for diabetes have been published by ADA/EASD [12] and AACE [13], with the purpose of providing guidance to healthcare providers caring for patients with type 2 diabetes and ensure best possible outcomes. Currently metformin is well accepted as the first line therapy for patients with type 2 diabetes in addition to lifestyle changes [2, 12-14]. There is no general agreement as to what is the best way to advance treatment in those who have not achieved target HbA1c levels with monotherapy [12, 13]. The current ADA and AACE guidelines both recommend an individualized approach to treatment intensification which should take into consideration cost, patient's preference, and profile of available medications [12, 13] It is generally accepted that patients with HbA1c level >10 % have a low probability of achieving ideal glycemic target of <7.0% with any of the traditional oral hypoglycemic agents, or even after basal insulin-only initiation. Therefore such patients will require prandial insulin, whether administered as a mixed formulation or basal-bolus regimen in order to archive glycemic goals [6, 12, 13, 15-26].

## 3. Insulin is a very effective glucose lowering agent, but it is associated with multiple side effects and shortcomings.

Patients with a very elevated HbA1c (>10%) are traditionally thought to have more advanced disease [2, 6] as well as glucotoxicity [27, 28], which coupled with the need to lower HbA1c by >3% to reach glycemic targets, make insulin an obvious treatment choice [15, 29]. Insulin is considered the most effective hypoglycemic agent and therefore capable of lowering HbA1c into target range regardless of baseline glycaemia [15]. Yet an insulin based treatment regimen, when implemented correctly and intensively, takes a significant toll on the patient's lifestyle by requiring a higher commitment to disease management in the form of more frequent self-monitoring, multiple daily injections, requires more frequent dose adjustments, and a greater investment in insulin-related diabetes education [30, 31]. Furthermore, insulin treatment

is commonly associated with two most undesirable side effects: weight gain and hypoglycemia [30, 32].

# 4. Treatment-induced weight gain has a negative effect on the disease pathophysiology and fuels its progression.

Most patients with diabetes are overweight and obese, development of which is often the initial event in the pathophysiology of type 2 diabetes [1, 33, 34]. Using therapeutic agents that focus primarily on blood glucose control but promote further weight gain seems counterintuitive, as this further worsens insulin resistance, which in turns results in an increase in insulin requirement, thus fueling a vicious cycle which promotes disease progression [35]. A Swedish study confirmed the deleterious effects of weight gain after diabetes diagnosis, as it demonstrated that patients with newly diagnosed diabetes who gain, rather than lose or maintain weight, are at a significantly increased risk of cardiovascular death [36].

# 5. Hypoglycemia is a common side effect of intensive insulin treatment and has far reaching consequences.

Hypoglycemia has a greatly underestimated effect on patients' life and beyond. Even seemingly minor hypoglycemic events create treatment related anxiety, heighten social anxiety, can limit or interfere with the patients' professional and social life, and can lead to treatment noncompliance. Hypoglycemia, especially severe hypoglycemia, has also been associated with untoward medical consequences like dementia, cardiovascular risk, seizures, and even death [30]. It also carries a great financial burden both in direct cost related to the event, as well as indirect costs like lost wages and work absenteeism [31]. The effects of hypoglycemia reach beyond the patient, affecting the psychological, social, and financial well-being of the whole family [37].

## 6. We need treatment algorithms which are patient-centric and offer the best overall benefit, rather than a glucose-centric approach.

With an ever increasing focus on personalized patient-centric treatment [12, 13], there is a renewed focus on patient-related outcomes, including treatment burden and quality of life. Insulin treatment requires an increased level of diabetes education, more intensive glycemic monitoring, a heightened awareness for potential side effects, a larger daily time commitment, all with potential negative effect on quality of life and treatment satisfaction [31, 37, 38]. The increase in treatment acuity related to insulin translates into higher healthcare related costs, a very timely concern for our economy [9-11, 31].

## 7. GLP-1 agonist have pleiotropic effects which target the core pathophysiologic abnormalities in type 2 diabetes.

- GLP-1 agonists have been a relatively recent addition to our diabetes treatment armamentarium. They exert many beneficiary actions, counteracting many of the basic pathophysiologic determinants of diabetes: enhance glucose stimulated insulin secretion, suppress glucagon production, promotes satiety, decreases food intake, improves insulin sensitivity, lower ectopic fat deposition (i.e. liver steatosis, visceral fat), etc. GLP-1
- agonists lower HbA1c by 1.5-2%, have a very low risk of hypoglycemia, and promote
- weight loss all very desirable effects in patients with type 2 diabetes [35]. While this

treatment does require an injection, it is very easy to use, does not require continuous treatment titration, and greatly reduces the need for frequent glucose self-monitoring. All these attributes make it quite an appealing treatment alternative for patients with type 2 diabetes. In the current diabetes treatment guidelines it is recommended as a second or third line agent after metformin failure.

8. The combination of basal insulin and GLP-1 agonists has been proven to be safe and very effective.

A meta-analysis of pooled data from across the LEAD program demonstrated that in patients with baseline HbA1c of > 9% liraglutide was better than glargine as an add on to oral hypoglycemic medications with average reduction in HbA1c of 1.9% [39]. Several other studies support equal or superior HbA1c reduction when a GLP-1 agonist is added to background therapy and compared to basal insulin, with the additional benefit of weight loss and minimal hypoglycemia [40-43]. GLP-1 agonist has also demonstrated superiority when added to maximized basal insulin therapy and metformin, when compared to prandial insulin alone [40, 44-48]. Furthermore, treatment with GLP-1 agonist in combination with basal insulin was shown to have a synergistic effect on glycemic control, with GLP-1 agonists exerting an insulin sparing effect, as well as ameliorating or eliminating the undesirable weigh gain associated with insulin therapy.

The current evidence suggests the combination of metformin, GLP-1 agonist, and basal insulin to be the most effective and simple strategy to achieve near normal glycemia in patients with a baseline HbA1c < 10%, while avoiding the side effects of weight gain, complexity of care, and hypoglycemia associated with insulin alone, or post-prandial hyperglycemia, weight gain, and hypoglycemia from the association of basal insulin to orals agents [40, 41, 43-48]. It is still not known whether these favorable effects extent to the more challenging group of patients with type 2 diabetes who have a baseline HbA1c >10%. Liraglutide reduces blood glucose by several mechanisms independent of insulin secretion and its superior effect on HbA1c and weight loss was found to be largely independent of diabetes duration and baseline HbA1c [39]. Treatment with GLP-1 agonists has also been associated with low secondary failure rates, durable and sustained long term blood glucose control, and durability of the initial weight loss [39, 42, 49].

Given all these distinct properties of GLP-1 agonists and simplicity of use, we propose they could represent a viable alternative to intensive insulinization in patients with very uncontrolled (HbA1c >10%) type 2 diabetes.

The aim of this study is to compare a GLP-1 plus basal insulin treatment regimen to a basal-bolus treatment regimen in patients with very uncontrolled (HbA1c>10%) type 2 diabetes. We will compare the two regimens with respect to efficacy in improving glycemic control, rate of hypoglycemia, change in weight, effect on patient quality of life, treatment burden, physician time, as well as healthcare related cost. We hypothesize that the two treatment regimens will have equal effectiveness, while the GLP-1 based regimen will be superior with respect to all other variables.

We chose to focus on a specific patient population which is generally considered to be most challenging to manage, use up greater heathcare resources, have higher potential for morbidity, and have traditionally been excluded from most clinical trials. Therefore this study will fill in an existing knowledge gap and provide high level evidence for future diabetes treatment guidelines pertaining to this patient population. We will obtain information not only in regards to the effectiveness of the treatment, but also safety and impact on healthcare cost beyond the cost of the drug.

Our findings will have great impact on the way we treat this – unfortunately – significant segment of the diabetic population, with huge potential benefits beyond just glycemic control, including quality of life, other metabolic co-morbidities, healthcare cost, etc. Additionally, if our proposed alternative regimen proves to be superior, this would represent a simple treatment alternative that primary care physicians can easily initiate and manage in their office, mitigating the need for referral to the specialist – representing a further healthcare cost control in addition to that observed in our study and a small step in alleviating the huge shortage of endocrinologists nationwide.

We are uniquely positioned to perform this study for multiple reasons: (1) we serve the largest county hospital in the US where this specific study population is greatly overrepresented; (2) our county hospital is a closed healthcare system, where all actual health-care related costs incurred by these patients can be readily captured; (3) the PI (and sub-I) have extensive clinical experience with this study population; (4) the PI has extensive clinical research experience, with proven track record of successfully designing clinically relevant studies and caring out to final completion even the most challenging research protocols.

## **SPECIFIC OBJECTIVES:**

We plan to evaluate a new GLP-1 based treatment strategy for patients with very uncontrolled (HbA1c>10%) type 2 diabetes and compare it to a standard basal-bolus insulin regimen.

Primary Specific Aim: To determine the non-inferiority of the basal insulin-GLP-1 agonist combination therapy to full basal-bolus insulin combination therapy in patients with very uncontrolled (HbA1c>10%) type 2 diabetes.

#### **Specific aims:**

- 1. Compare the two treatment regimens with respect to a disease and patient-relevant composite outcome of effectiveness (HbA1c <7%) and safety (no hypoglycemia and no weight gain);
- 2. Compare the two treatment regimens with respect to treatment burden (number of daily shots, amount of glucose self-monitoring, need for treatment titration);
- 3. Compare the two treatment regimens with respect to quality of life [as measured by a disease specific (DQOL) questionnaire and general heath (SF-36) questionnaire];

4. Compare the two treatment regimens with respect to all healthcare related costs: actual cost of the pharmacologic agents, glucose monitoring supplies, all other pharmacologic (non-study related) and non-pharmacologic healthcare related costs (outpatient and inpatient, diabetes related and non-diabetes related). We will also compare actual physician time spent during office visits and non-visit related care of these patients. While no actual dollar amount can be attached to this (phone visits and longer office visits required by the need for extra patient education are not customarily reimbursable) time commitment is of great relevance to our physicians who care for these very complex patients.

Primary outcome:

220

221

222

223

224

225

226

227

228

229230

231

232233

234

235

236

237

238

239

240

241

242

243

244

245

246

247

250

Change in HbA1c from randomization to 26 weeks of therapy.

**Secondary outcomes:** 

- 1. The main secondary outcome is a less traditional but very patient-centric and clinically meaningful composite outcome of HbA1c <7% AND no documented hypoglycemia (capillary glucose level <56 mg/dl) AND no significant weight gain (<3% body weight) during the 6-mo study follow-up;
- 2. % reaching target HbA1c of <7% at end of study;
- 3. 7-point glucose profile results;
- 4. % patients reaching pre-specified "treatment failure" outcome;
- 5. Change in weight from baseline (both absolute weight lost and percent of body weight);
- 6. % patients with weight loss >5% of body weight;
- 7. Number of hypoglycemic episodes defined as mild (symptoms of hypoglycemia confirmed by a CBG reading of <70 mg/dl), moderate (any CBG reading <56 mg/dl), severe (need for help to recover regardless of CBG reading);
- 8. Number of patients experiencing any hypoglycemic episodes;
- 9. DQOL questionnaire score;
- 249 10. SF-36 questionnaire score;
  - 11. Number of daily injections;
- 251 12. Total daily dose of insulin;
- 252 13. Health care cost, total:
- 253 14. Health care cost, diabetes-related;
- 254 15. Total number of CBG checks/study;
- 255 16. Number of CBG checks/month;
- 256 17. Number of titration events by healthcare professional;
- 257 18. Number of titration events by patient;
- 258 19. Healthcare provider time during scheduled office (minutes/visit);
- 259 20. Healthcare provider time, unscheduled (total minutes);
- 260 21. Compliance with pharmacologic therapy;
- 261 22. Change in LDL cholesterol from baseline;
- 262 23. Change in Triglycerides from baseline;
- 24. Tolerability defined as percentage of patients with side effects (other than hypoglycemia) related to the study medications;

25. Tolerability - defined by percentage of patients dropping out of the study due to side effects related to the study medications.

267 268 269

270

271

272

273

274 275

265

266

## RESEARCH DESIGN AND METHODS

## **Study type:**

- Single Center (UT Southwestern Medical Center at Dallas, TX)
- Randomized
- Single blind (evaluator)
  - Two treatment arms (treatment and control)
  - Length of intervention: 6 months
  - Efficacy & safety trial
  - Non-inferiority trial for primary outcome

277 278 279

276

## **Study Design:**

280 We will conduct a prospective, randomized, single blind, two-arm, parallel trial 281

comparing two treatment regimens (liraglutide, detemir, and metformin versus aspart,

detemir, and metformin) in patients with very uncontrolled (HbA1c>10%) type 2 282

283 diabetes. The investigator performing the study related measurements will be blinded to

284 the patients' treatment assignment.



286 287

Figure 1: Study design showing the run-in period, followed by the randomization visit and the 6-mo intervention period.

288 289 290

291

The University of Texas Southwestern Medical Center Institutional Review Board will review the study and approve all relevant documents. Furthermore, study approval will be obtained from Parkland Health and Hospital System (PHHS), which represents the study site.

294 295

292

293

296

297

298

299

300 301

302

303

304

305

### **Rationale for study Design**

- The randomized design, with stratification for pertinent variables, will allow us to fully compare the effects of the two treatment algorithms in this hard to treat patient population.
- A 3-7 day run-in period was introduced in order to ensure patient compliance with study procedures prior to randomization.
- The patient-guided titration schedule for basal insulin is well validated in the literature and should help to lower fasting glucose level within a shorter period of time.
- A 6-month intervention period was chosen as nadir HbA1c after initiation of a treatment regimen is achieved by this time, therefore allowing us to evaluate the full effectiveness of these interventions.

306 307 308

#### **Study Population:**

309 Inclusion Criteria:

- 310 1. Informed consent obtained before any trial-related activities;
- 311 2. Both genders and all ethnicities;
- 312 3. Currently receiving medical care at Parkland Health and Hospital System (PHHS),
- 313 Dallas, TX;
- 314 3. Age > 18 years;
- 315 4. Diagnosis of Type-2 Diabetes, regardless of time since diagnosis;
- 5. Confirmed HbA1c > 10%. 316

317 318 319

320

321

322

323

324

325

326 327

328

329

330

331

332 333

334

335 336

#### Exclusion criteria:

- 1. Age <18 as the feasibility and safety of this treatment regimen should be first established in the adult population; if successful, a subsequent pediatric study will be proposed:
- 2. Current use (within the past 30 days) of prandial-insulin;
- 3. Current use (within the past 30 days) of GLP-1 analogues or DPP-4 inhibitors;
- 4. Type 1 diabetes as purposefully withholding meal-time insulin is contraindicated;
  - 5. Clinical state requiring inpatient admission/treatment;
  - 6. Contraindication or strong cautions to any of the study medications:
    - a. eGFR <30 ml/min if already on metformin, or eGFR<45 ml/min is not currently on metformin (per metformin label)
    - b. History of lactic acidosis (per metformin label)
    - c. Advanced hepatic or cardiac disease (per metformin label)
      - d. Age >80 years (per metformin label)
      - e. Chronic alcohol use (>14 drinks/week)
      - f. History of pancreatitis (per liraglutide label)
- g. Personal or family history of medullary thyroid cancer or MEN syndrome (per liraglutide label)

- h. Pregnancy, intention of becoming pregnant, or lactation (per liraglutide label)
  - i. Female of reproductive age not using adequate contraceptive methods (per liraglutide label). Adequate contraceptive measures include sterilization, intrauterine devices, oral contraceptives, approved hormonal implant, diaphragm with spermicide or condom with spermicide;
  - 7. Any serious or unstable medical condition as it would interfere with treatment assignment as well as outcome measurement;
  - 8. Any scheduled elective procedures/surgeries;
  - 9. Active infections, including osteomyelitis;
  - 10. Not willing to participate, unable to keep projected appointments, unwillingness to receive injectable treatment;
  - 11. Known or suspected allergy to any of the trial products or related products;
  - 12. Prior participation in this or another trial, or receipt of any investigational drugs within 3 months prior to screening;
  - 13. Non-English speaking patients are excluded for safety reasons.

353354 Rationale for Study Population

Patients who have a very elevated HbA1c (>10%) are thought to have significant glucose and lipotoxicity and the current guidelines recommend initiation of a full insulin regimen. This is a difficult to treat population, as they generally have more advanced disease, less beta-cell reserve, and, often time, poor compliance. Finding a simpler, safer, and effective treatment algorithm for these patients would have a great impact on the rate of comorbidities, as well as healthcare cost. This is also a population traditionally excluded from all regulatory studies, therefore little information is available on how to best approach their treatment.

**Rationale for Study Location** 

Only patients from the PHHS system will be recruited. PHHS is a county hospital that provides comprehensive care (primary, specialty, inpatient and outpatient) to the indigent population of Dallas County. EPIC is the electronic medical record that is deployed at all sites and covers all aspects of care, including financial data. Therefore PHHS is the ideal location to conduct this study, as all patient-related information is captured and can be queried at multiple levels, including cost.

**Randomization Criteria** 

1. Patient returned a fully completed 7-point glucose profile – suggesting likely compliance with proposed study procedures.

Withdrawal Criteria

- 1. The subject may withdraw consent at any time.
- 2. Severe drug-related side effects including (but not limited to) acute pancreatitis, severe nausea and/or vomiting, renal failure, diagnosis of medullary thyroid cancer, or hypersensitive to any study drug.
- 3. Pregnancy or intention of becoming pregnant.
- 4. Subject's diabetes control remains unchanged or becomes worse.

- 5. Subject participation in the research is no longer safe
  - 6. The researchers believe that other treatment may be more helpful.
- 7. The sponsor or the FDA stops the research for the safety of the participants.
  - 8. The sponsor cancels the research.
    - 9. Subject is unable to keep appointments or to follow the researcher's instructions.

## **Subject Replacement**

Subjects who withdraw or become ineligible will not be replaced. A drop-out rate of 12% is estimated and already calculated in the recruitment plan.

#### **Study Schedule**

394 Recruitment:

We will recruit patients from the following locations within the PHHS: emergency room (only if discharged home after the evaluation), primary care clinics, any specialty clinic (including diabetes clinic). Eligible patients will be informed about the trial by their treating physician. If agreeable, they will be contacted by the study staff and a screening appointment scheduled as soon as feasible (within days).

Screening Visit (visit 1):

During the screening visit patients will complete the informed consent process and will undergo a complete assessment for all inclusion and exclusion criteria. A complete medical history and comprehensive physical examination will be performed. Blood will be drawn (if not done within the past 7 days) to assess for all eligibility criteria (HbA1c, creatinine, liver function tests and pregnancy test, if applicable). Patients will receive an identification card with information about participation in the study. Patients will be asked to complete a 7-point glucose profile on the day prior to their next visit.

Randomization (visit 2):

Randomization will occur at the second visit (3-7 days from visit 1-screening). The study statistician will generate a blocked randomization scheme (1:1) stratified by "any insulin treatment at time of screening" (yes/no) and BMI (cutoff 37 kg/m2 – the average BMI of this study population in our PHHS Diabetes Clinic).

At this visit we will obtain a full baseline evaluation of all outcome parameters. All patients will meet with the dietician to received education regarding recommended lifestyle modifications. Patient will undergo diabetes education as well as teaching regarding insulin injection and titration.

- *Phone follow-up/ Drug titration visit:*
- At 2-wk from randomization (visit 3) a phone visit will take place to assess for safety parameters (particularly hypoglycemia) and perform protocol-driven treatment titration.

- 425 Follow-up visits:
- At 1-, 3-, and 6-months (visits 4, 5, 6) patients will be followed-up in person for interim
- 427 (and end of study, respectively) evaluations of all outcome parameters, as well as

protocol-driven treatment titration. A 7-point glucose profile will be repeated prior to the last visit in the study.

431 Interventions:

 Both groups will either continue or initiate treatment with metformin. To minimize gastrointestinal side effects metformin will be initiated at 500 mg daily (or continued at current dose) and titrated weekly in 500 mg increments to the final dose of 1000 mg twice daily (or maximum tolerated dose which should be at least 500 mg BID).

Both groups will be initiated on basal insulin detemir. If new to insulin, this will be started at 0.3 units/kg once daily at bedtime and self-titrated based on the study protocol (see detemir patient self-titration table). If already on basal insulin, will take the total daily dose of basal insulin and perform a 1:1 dose conversion to insulin detemir, which will be administered once daily at bedtime, followed by the same titration. Additionally, physician-directed titration will occur, if needed, during the scheduled phone and/or office visits, as well as any unscheduled patient-initiated visits (phone/in person, if applicable). All patients new to insulin will be seen by the diabetes educator to receive instruction in insulin injection techniques.

Detemir patient self-titration table:

| Fasting Blood glucose | Change in your insulin dose |
|-----------------------|--------------------------------|
| <45 | Decrease by 5 units |
| <70 mg/dL | Decrease by 3 units |
| 71- 100 mg/dL | No change in your insulin dose |
| 101-120 mg/dL | Increase by 1 units |

Patients randomized to liraglutide will stop any insulin products besides detemir (if applicable), initiate liraglutide at 0.6 mg/day, and dose escalate weekly to 1.2 mg/dl and final dose of 1.8 mg/dl. Patients who develop significant and persistent gastrointestinal side effects are allowed to down-titrate the dose of liraglutide to 1.2 mg/dl for 1 week or until the side effect resolve.

Patients randomized to meal-time insulin will initiate insulin aspart before each meal. Aspart insulin will be initiated at a dose of 0.3 units/kg/day divided among the number of meals taken daily. Meal-time insulin titration, if needed, can be either patient driven (see table below) or physician-directed during the scheduled follow-up visits (phone or in person), as well as any unscheduled patient-initiated visits (if applicable).

Novolog patient self-titration table:

| Novolog patient sen-titration table. | | | | | |
|---|---|---|---|---|---|
| Glucose | Change in | Glucose | Change in | Glucose | Change in |
| prior to | breakfast | prior to lunch insuli | | prior to | dinner |
| lunch | insulin dose | dinner | dose | bedtime | insulin dose |
| <54 | -2 units | <54 | -2 units | <54 | -2 units |
| 55-69 | -1 unit | 55-69 | -1 unit | 55-69 | -1 unit |
| 70-120 | No change 70-120 | | No change | 70-130 | No change |
| 121-160 | +1 unit | 121-160 | +1 unit | 131-180 | +1 unit |

| >160 | +2 units | >160 | +2 units | >180 | +2 units |
|------|----------|------|----------|------|----------|

## **Rescue therapy:**

Should any patients randomized to liraglutide treatment experience persistent hyperglycemia (defined as a confirmed Hb1c>10%) at the 3-mo visit (visit 5), meal-time insulin aspart will be initiated per the same protocol as above. This is a pre-specified "treatment failure" end-point. Following initiation of rescue therapy patients will continue all scheduled visits and procedures through the end of the trial.

Should any patients randomized to the "standard of care" group experience persistent hyperglycemia (defined as a confirmed HbA1c >10%) at the 3-mo visit (visit 5), treatment and insulin titration will continue as scheduled. This is also a pre-specified "treatment failure" end-point.

475 A graphical review of the visit procedures and timing is presented below:

| 8 1 | 5 1 | | | | | |
|---|---|---|---|---|---|---|
| Visit | 1 | 2 | 3 | 4 | 5 | 6 |
| | 3-7 | | | 1 | 3 | 6 |
| Time | days | 0 | 2 weeks | month | months | months |
| Type | Office | Office | Phone | Office | Office | Office |
| Consent | X | | | | | |
| I&E criteria | X | | | | | |
| Randomization criteria | | X | | | | |
| Randomization | | X | | | | |
| Physical exam | X | | | X | X | X |
| Height | X | | | | | |
| Vitals (weight, BP, pulse) | X | X | | X | X | X |
| Dietary counseling | X | X | X | X | X | X |
| Lifestyle counseling | X | X | X | X | X | X |
| 7-point glucose | | X | | | | X |
| Labs (HbA1c, lipids, CMP, Hb) | X | | | | X | X |
| Dispense trial drug | | X | | X | X | |
| Hypoglycemia assessment | X | X | X | X | X | X |
| Frequency of glucose monitoring | | | | X | X | X |
| Titrate insulin | | X | X | X | X | |
| Liraglutide titration (if applicable) | | | X | | | |
| Insulin dose assessment | | X | X | X | X | X |
| Compliance assessment | | | | X | X | X |
| # daily injections | | | | X | X | X |
| QoL questionnaires (DQOL and | | | | | | |
| SF36) | | X | | | | X |
| AE and SAE assessment | | X | X | X | X | X |
| Pregnancy test (if needed) | X | X | | X | X | X |
| Physician time assessment | | X | X | X | X | X |
| Healthcare cost data extraction | | | | | | X |

### Dietary Modifications:

Counseling regarding the type and amount of food consumed with strong encouragement to count carbohydrates and/or calories will be performed for all patients by the dietitian at visit 2 and investigator at visits 3-5.

## <u>Lifestyle Modifications:</u>

All patients will receive recommendations regarding type/amount/intensity of physical activity and be provided future goals at visit 1. Reinforcement of these objectives will take place at visits 2-5.

#### **Assessments for Efficacy**

- 1. <u>HbA1c</u> measured at screening, visit 5 (3-months) and end of study (6 months). Samples are processed immediately and stored at 0-5°C. It will be analysed within 24 hrs at the UT Southwestern Medical Centre Diabetes laboratory using an HPLC technique. The laboratory is accredited by the National Glycohemoglobin Standardization Program. HbA1c interassay coefficient of variability is ≤2%, and the intra-assay variability is ≤0.3%.
- 494 2. Weight will be measured at each office visit using the same calibrated digital scale, while patients wearing no shoes and only light clothing.
- 496 3. Total daily insulin dose will be calculated in units/kg at each visit by summing all insulin shots of all types over a 24 hrs period. The average of the 3 most recent 24 hrs prior to each visit will be used.
  - 4. <u>Number of daily injections</u> will be counted at each visit, by adding all shots regardless of the type of insulin. The average of the 3 most recent 24 hrs prior to each visit will be used.
- 502 5. Systolic and diastolic blood pressure will be measured in sitting position using an Omron digital manometer, on the right arm, after 5 minutes of rest.
  - 6. <u>Lipid profile, liver function test, haemoglobin will</u> be collected at screening, 3-months, and end of study in fasting state. The blood will be processed and analysed immediately by PHHS Clinical Laboratory.
  - 7. <u>7-point glucose measurement</u> will be performed by the patient on the day prior to the randomization visit and prior to the end-of-study visit.
  - 8. <u>Frequency of glucose monitoring</u> will be assessed by downloading the glucose monitor. Average number of readings/day will be recorded at each visit.

#### **Assessments for Safety**

All safety assessments are performed at each visit, in person or by phone. Any unanticipated or serious adverse events will be reported to the local IRB and FDA in accordance with local guidelines.

- 1. <u>Hypoglycemia</u> All plasma glucose values ≤ 70 mg/dL, as well as values >70 mg/dL when hypoglycemic symptoms have occurred, should be recorded by the subjects in the blood glucose diaries provided at each visit. The recording should include:
- date of hypoglycemic episode

- time of hypoglycemic episode
- time of last main meal prior to episode
- whether the episode was symptomatic
- whether the episode was in relation to exercise
- whether seizure or coma developed
  - whether the subject was able to treat him/herself
  - the plasma glucose level before treating the episode

531

532

533

534

535

536

537

538

539

540

541

542

527

- The following definitions for hypoglycemia will be used:
  - Mild- Symptomatic or asymptomatic hypoglycemia with blood glucose 56-69 mg/dl and subject was able to treat him/herself
  - Moderate- Symptomatic or asymptomatic hypoglycemia with blood glucose <56 mg/dl and subject was able to treat him/herself</li>
    - Severe- Blood sugar <70 mg/dl or symptoms highly suggestive of hypoglycemia and the subject needed assistance to be treated with carbohydrates, glucagon, or other resuscitative actions
    - Nocturnal hypoglycaemia- blood glucose <70 with a time of onset between 00:01 and 05:59 (both included)
    - Relative Hypoglycemia- Blood glucose >69 mg/dl with symptoms highly suggestive of hypoglycemia
    - Probable symptomatic hypoglycemia- Symptoms highly suggestive of hypoglycemia but subject did not measure blood glucose.

543544545

546

547

548

549

550

551

552

553

- 2. Other treatment specific side effects
  - Nausea, vomiting, diarrhea, and headache;
  - Abdominal pain suspicious for pancreatitis would prompt immediate physician evaluation and laboratory testing for amylase and lipase measurement which would be processed immediately and analysed by PHHS Clinical Laboratory.

3. <u>Pregnancy Test</u>- females of childbearing potential will have urine pregnancy test (human chorionic gonadotropin, hCG) performed if clinically indicated in the assessment of the investigator. Urine-stick pregnancy test will be performed for females of childbearing potential at any time during the trial, if a menstrual period is missed or if the participant voices concern.

554555556

#### Other Assessments

557 <u>Treatment satisfaction and quality of life</u> will be assessed at the randomization visit (Visit 558 2) and end of study (Visit 6) using a modified DQoL and SF-36 questionnaires. Total score as well as individual domain scores will be analysed and reported.

- 561 <u>Subject Compliance:</u> Participants will bring all study medication to each appointment for
- review and study drug will be distributed at each appointment (visit 1, 2, 3, 4, and 5).
- Percent compliance will be calculated and recorded at each visit.

<u>Healthcare Cost Assessment:</u> At the conclusion of the study, the EPIC integrated medical record system will be queried for the data regarding all healthcare related expenditures. From this information a data subset of diabetes-related expenditure will also be reported.

<u>Physician Time Assessment:</u> Each physician interaction (office visit or phone visit) will be timed to compare the two treatment regimens with respect to burden on healthcare provider's time.

## RISKS ASSOCIATED WITH THE PARTICIPATION IN THE STUDY: Risks of Liraglutide:

Very common (reported by more than 10 percent of the patients):

 Gastrointestinal adverse events are the most common side effect of liraglutide and reported in up to 41% of patients. Nausea is seen in approximately 13% of patients treated with liraglutide and is usually developed in the first 2 weeks. It tends to be mild, dose-related and decline over time. In some patients the nausea can be more severe and be associated with vomiting which is usually transient and self-resolving.

Common (reported by 5-10 percent of the patients)

Low blood sugar (hypoglycemia) - - The risk of having hypoglycemia with liraglutide is higher if taking it with another medicine that can cause hypoglycemia, such as a sulfonylurea or insulin. In some people, the blood glucose may get so low that they need another person to help them. The dose of your sulfonylurea medicine or insulin may need to be lowered while using liraglutide.

• Headache and upper respiratory tract infections have been reported in 7-9% of patients treated with liraglutide. A similar percentage of patients developed headaches with placebo or comparator drug.

Uncommon side effects (reported by 1-5 percent of the patients):

Injection site reactions (e.g., injection site rash, erythema) were reported in approximately 2% of liraglutide treated patients in the five clinical trials of at least 26 weeks duration. Less than 0.2% of liraglutide-treated patients discontinued due to injection site reactions.

Very rare side effects (affects less than 1 percent of patients)

Acute pancreatitis (inflammation of the pancreas) - there have been few reported event of acute pancreatitis presenting with persistent severe abdominal pain (usually accompanied by vomiting). Patients experiencing the above symptoms should contact the study doctor who will decide on whether they should discontinue the trial medication and /or require additional diagnostic procedures.

• Rarely, a severe form of allergic reaction (anaphylactic reaction) with additional symptoms such as breathing problems, swelling of throat and face, fast heart beat

- etc. has been reported with marketed use of Liraglutide. Patients experiencing these symptoms should seek immediate medical help and inform the trial doctor as soon as possible.
  - Kidney failure Liraglutide may cause nausea, vomiting or diarrhea, leading to loss of fluids (dehydration). Dehydration may cause kidney failure which can lead to the need for dialysis. This can happen in people who have never had kidney problems before. Drinking plenty of fluids may reduce the risk of dehydration.

## Other potential risks related to liraglutide:

- Hyperglycemia (too high blood glucose) can occur, especially if there is insufficient treatment. The symptoms of hyperglycemia include increased urination, feeling thirsty, losing appetite, feeling sick (nausea or vomiting), feeling drowsy or tired, flushed, dry skin, dry mouth and a fruity (acetone) smell of the breath. If not treated, these symptoms may develop into a serious condition called diabetic ketoacidosis which may even lead to death.
- Thyroid tumors, including cancer -During the drug testing process, the medicine in Victoza caused rats and mice to develop tumors of the thyroid gland. Some of these tumors were cancers. It is not known if Victoza will cause thyroid tumors or a type of thyroid cancer called medullary thyroid cancer in people. If medullary thyroid cancer occurs, it may lead to death if not detected and treated early. If you develop tumors or cancer of the thyroid, your thyroid may have to be surgically removed. Fibrosarcomas (cancer underneath the skin) were seen at the point of injection (skin) in male mice that underwent a 2 year study of liraglutide. These fibrosarcomas were attributed to the high local concentration of drug near the injection site. The liraglutide concentration in the preparation used for humans is 10 times higher than the concentration used in mice. It is not known if liraglutide will cause fibrosarcomas in people.

## Risk of insulin detemir and aspart:

## Very common (1-10 in 100 patients):

- Hypoglycemia (low blood sugar) is the most common adverse reaction of insulin therapy and may be life- threatening if severe and not treated appropriately.
- Mild-moderate weight gain is expected with any insulin therapy

## Less common (less than 1 in 100 patients):

- Severe, life-threatening, generalized allergy, including anaphylaxis, can occur with any insulin products, including detemir insulin or aspart insulin.
- Other adverse reactions associated with detemir insulin and/or aspart insulin include injection site reactions, lipohypertrophy, rash, itching.
- Needles and insulin pens should never be shared.

#### Risk of Metformin:

Very common (1-10 in 100 patients):

- 656 Abdominal or stomach discomfort
- Decreased appetite
- 658 Diarrhea
- Bloating

• Low serum Vitamin B12 levels without clinical manifestations

## Precautions:

- Lactic Acidosis: Lactic acidosis is a very rare, but serious, metabolic complication that can occur due to Metformin accumulation during treatment with Metformin HCl; when it occurs, it is fatal in approximately 50% of cases. Lactic acidosis may also occur in association with a number of pathophysiologic conditions, including diabetes mellitus. Metformin should be discontinued immediately and health care provider should be promptly notifed if unexplained increase in breathing rate, muscle aches, fatigue and unusual somnolence occur.
- Patients with Renal disease or renal dysfunction (e.g., as suggested by eGRF <30 ml/min) should not use metformin</li>
- Metformin should be temporarily discontinued 48h prior to radiologic studies involving intravascular administration of iodinated contrast materials 48h prior to procedure to avoid increased risk of development of lactic acidosis and restarted 24h after the procedure.
- Excessive alcohol intake, either acute or chronic should be avoided while receiving Metformin.

## SAFEGUARDS AND PRECAUTIONS TO MINIMIZE RISKS/HARMS:

- Hypoglycaemia episodes will very closely monitored trough the study using self-glucose monitoring. Review of blood glucose diary and hypoglycaemic events will be discussed during office, phone visits and as needed. Patient will be instructed during randomization visit on how to proper handle mild, moderate and severe hypoglycemic episodes and how to reduce their basal insulin doses according to study protocol. Those instructions will be reinforced as needed during the study.
- Should any patients randomized to liraglutide treatment experience persistent hyperglycemia (defined as Hb1c>10%) at the 3-mo visit (visit 5), meal-time insulin aspart will be initiated per the same protocol as the standard group
- Should any patients randomized to the "standard of care" group experience persistent hyperglycemia (defined as HbA1c>10%) at the 3-mo visit (visit 5), treatment and insulin titration will continue as scheduled.
- Patients will be monitored closely for any drug-related side effects. They will be provided with instruction on when to call the PI and a direct phone line, so they can immediately report any problems or concerns. Instructions will be given on possible side effects and how to avert/minimize them.

• Only qualified personnel will perform blood draws to minimize the risk of complications.

• Patients are allowed to skip questions on the questionnaire should they feel that the question might pose a psychological burden.

## STATISTICAL CONSIDERATIONS:

## **Sample Size Calculation**

We propose to test a non-inferiority hypothesis comparing the 6-month change from baseline in HbA1c between the two treatment groups, with a non-inferiority margin of 0.4%. We conservatively estimate the standard deviation of the difference at 0.5% based on results from reported studies with similar design[44, 45, 47]. Using a one-sided alpha of 0.025, we determine that 44 subjects per group completing 6 months will provide power 0.96 to test this non-inferiority hypothesis, shown below amongst with other scenarios (Hintze, J. (2011). PASS 11. NCSS, LLC. Kaysville, Utah, USA. <a href="https://www.ncss.com">www.ncss.com</a>). We will need to randomize 100 patients to test this hypothesis assuming a 12% drop-out rate (estimated drop-out rate based on our extensive prior experience with similar population and length of study). We plan to screen 120 patients to account for approximately 20% anticipated screen failures.

Power and sample size estimation for Non-Inferiority Test (H0: Diff >= NIM;

H1: Diff < NIM)

Higher Means are Worse Test Statistic: T-Test

| | | Non- | | | | |
|-------|-------|-------------|------------|--------------|-------|------------|
| | | Inferiority | Actual | Significance | | Standard |
| | | Margin | Difference | Level | | Deviation1 |
| Power | N1/N2 | (NIM) | (D) | (Alpha) | Beta | (SD1) |
| 1.000 | 44/44 | 0.4 | 0 | 0.025 | 0.000 | 0.3 |
| 1.000 | 48/48 | 0.4 | 0 | 0.025 | 0.000 | 0.3 |
| 1.000 | 50/50 | 0.4 | 0 | 0.025 | 0.000 | 0.3 |
| 0.960 | 44/44 | 0.4 | 0 | 0.025 | 0.040 | 0.5 |
| 0.973 | 48/48 | 0.4 | 0 | 0.025 | 0.028 | 0.5 |
| 0.977 | 50/50 | 0.4 | 0 | 0.025 | 0.023 | 0.5 |
| 0.755 | 44/44 | 0.4 | 0 | 0.025 | 0.245 | 0.7 |
| 0.791 | 48/48 | 0.4 | 0 | 0.025 | 0.209 | 0.7 |
| 0.808 | 50/50 | 0.4 | 0 | 0.025 | 0.192 | 0.7 |

Further, this sample size will yield at least 80% power at two-sided alpha=0.05, superiority hypothesis, for the secondary composite outcome endpoint of HbA1c<7% with no hypoglycemia and no significant weight gain, expecting that 25% and 5% reach

this endpoint with liraglutide treatment and standard basal-bolus insulin treatment, respectively.

727 728 729

730

731

732

726

#### Randomization

Treatment assignment will occur at the second visit. The study statistician will generate a blocked randomization scheme (1:1) stratified by "any insulin treatment at time of screening" (yes/no) and BMI (cutoff 37 kg/m2 – the average BMI of this study population in our PHHS Diabetes Clinic), programmed using SAS Proc Plan.

733 734 735

736

737

738

739

740

741

742

743

744

745

### Statistical Analysis Plan

All statistical analyses will be performed by the study statistician (Beverley Huet), who has extensive experience in clinical trials analysis.

Primary analysis: The primary analysis will be intention-to-treat (ITT) which will include all randomized participants who receive at least one dose of a study medication. The non-inferiority of liraglutide treatment strategy compared to standard basal-bolus insulin regimen will be assessed using a 95% confidence interval for the between treatment group net difference (month 6 minus month 0) in HbA1c at 6 months. This 95% confidence interval will be derived from the differences of least square means estimated from a mixed model repeated measures analysis. Non-inferiority of liraglutide treatment will be concluded if the upper limit of the 95% confidence interval is less than the non-inferiority margin of 0.4%.

746 747

748 Secondary analyses: We will also perform a per-protocol analysis comparing HbA1c 749 response because, in non-inferiority hypothesis testing, the ITT analysis may be biased 750 toward the null hypothesis. The per-protocol population is defined as the population who 751 continued the assigned intervention as randomized for the duration of the study period. 752 Secondary outcomes include the composite endpoint of HbA1c<7% with no 753 hypoglycemia and no significant weight gain, a binary variable, which will be compared 754 between the randomized study groups with a logistic regression model. The odds ratio 755 and corresponding 95% confidence intervals will be reported. From healthcare related 756 cost data, cost-effectiveness ratios will be summarized as point estimates with 95% 757 confidence intervals, accounting for the skewness in the distribution of the ratio [50]. 758 Sensitivity cost analyses will be performed to further assess variables such as treatment 759 failure and quality of life weights. Multiple logistic regression models will be constructed 760 to evaluate any association of baseline covariates on treatment efficacy. Binary 761 secondary endpoints will also be assessed with logistic regression models. Group 762 comparisons and changes from baseline over time (study visits) of continuous secondary 763 outcome variables will be analysed with mixed model repeated analysis. The logrank test 764 will be used to compare the pre-specified "treatment failure" end-point between groups. 765 Safety endpoints and hypoglycemic and other adverse events will summarize in detail 766 with descriptive statistics. The analysis of safety data will be performed for the ITT 767 population.

Model assumptions regarding normality and covariance structure will be carefully assessed. Nonparametric tests or data transformations will be used if necessary to meet assumptions. Statistical analysis will be performed with SAS software (SAS Institute, Cary NC), particularly Proc Mixed for linear models with both fixed and random effects.

772 A two-sided alpha <5% will be considered significant for all analyses.

## **Interim Analysis**

No interim analysis is planned.

## **DATA HANDLING AND RECORD KEEPING:**

All data will be collected in strict compliance with the University's HIPPA rules. Research records (source documents) will be kept in a double-locked filing system in a secure locked room. Collected data will be stored in an electronic study database will be encrypted and password protected and saved on the University's secure network. Only study personnel will have access to these records.

The institutional review board (IRB) governing this study may inspect the medical records of any patient involved in this study at any time.

Laboratory specimens will be collected under standard of care protocol at Parkland hospital laboratory and handled in accordance with the hospital policy.

The study blind will be maintained by the designated statistician and only broken by request from a treating physician in case of a medical emergency.

#### **ETHICS:**

**Ethical Considerations:** 

- 1. Exclusion of non-English speakers- while translators are available during working hours, the investigators are worried that no translator will be available to assure safety measures at all times.
- 2. Compliance with Insulin Regimen- At times patients are not compliant with complicated insulin regimens and providers often continue to uptitrate insulin dosage when patients remain above HbA1c goal. If patient compliance improves once enrolled in the study, there is a higher risk of hypoglycemia. Every effort will be made at all visits to determine exactly what amount of insulin the patient is taking and the overall compliance.

## **Informed Consent:**

Informed consent will be obtained during the first face-to-face contact. Once a prospective subject is identified, we will explain the study details and preliminary eligibility is accessed either through phone or face-to-face interview. If the prospective volunteer remains interested in the study and fulfils preliminary eligibility criteria, baseline studies are scheduled. Only study personnel listed on the consent will be permitted to obtain consent. The subject will be provided informed consent and it will be signed and witnessed. The consent form will discuss the procedures to be performed at each visit, the number of visits, and what is expected of the patient, along with all possible side effects. A copy will be given to the subject and the original will be kept on file. Potential subjects may be screened for eligibility using a study-specific HIPAA waiver. Volunteers who call to inquire about the study will have their demographic and contact information collected over the phone, and the study will be described to them.

- 818 Once the subject has agreed to participate and appears in person, a study specific HIPAA 819 Authorization will be signed, along with the consent form document. 820 821 Confidentiality/HIPAA: 822 Every effort will be made to keep all information about the patient confidential. Consent 823 forms will be placed in the patient charts. Research records will be kept in a double-824 locked filing system in a secure locked room. The electronic study database will be 825 encrypted and password protected and saved on the University's secure network. Only 826 study personnel will have access to these records. 827 828 The institutional review board (IRB) governing this study may inspect the medical 829 records of any patient involved in this study. 830 831 IRB Approval: 832 The study is approved by the UT Southwestern IRB. 833 834 FDA Approval: 835 An IND/NDA exception was granted by the FDA for possible use of rescue therapy with 836 prandial insulin add-on to detemir-liraglutide combination should patients in the 837 liraglutide arm reach the pre-defined failure end-point. 838 839 Declarations: 840 This study will be conducted in accordance with the Declaration of Helsinki. This study will be conducted in accordance with the ICH GCP guidelines. 841 842 The sponsor-investigator will comply with all applicable regulatory and legal 843 requirements, ICH GCP guidelines, and the Declaration of Helsinki in obtaining and 844 documenting informed consent. 845 846 Study schedule: IRB approval: December 2013 847 848 Start of Study: as soon as funding received (estimate March 2014) 849 Recruitment period: March 2014 – February 2015 850 First Patient First Visit: March 2014 851 Last Patient First Visit: February 2015 852 Last Patient Last Visit: August 2015 Final Report: October 2015 853 854 Final Manuscripts: December 2015 855 856 **STUDY DRUGS AND MATERIALS:** 857 **Study medication**
- 858 Liraglutide 6 mg/ml solution for subcutaneous injection delivered in a 3 ml prefilled
- disposable pen

- 860 Detemir insulin 300 units/prefilled disposable pen
- Aspart insulin 300 units/prefilled disposable pen

Provided and manufactured by NovoNordisk A/S.

864 865 NovoFine Pen needles – provided by NovoNordisk US. 866 867 Storage and Drug Accountability of Study Medication(s) Patients will be instructed as follows: 868 869 -Store unused pens in a refrigerator at a temperature between +2°C and +8°C 870 (36°F to 46°F). Keep away from the cooling element. Do not freeze and do not 871 use if it has been frozen. 872 -Store pens in use for 30 days at room temperature (15°C to 30°C; 59°F to 86°F) 873 or in a refrigerator (2°C-8°C; 36°F to 46°F). 874 -Do not freeze and do not use if it has been frozen. 875 -The pen must be protected from all sources of light, and the pen cap should be 876 kept on when the pen is not in use. -Product should not be used if it does not appear clear and colorless. 877 878 Investigator will ensure availability of proper storage conditions and record and evaluate 879 the temperature. While at the site, drug will be stored in a temperature-monitored 880 refrigerator at 4°C. 881 There will be no trial medication dispensed to any person not enrolled in the study. 882 Unused medication will be stored separately from used trial medication(s). 883 Procedures for Drug Accountability: 884 -At study site all trial products will be kept in locked refrigerator and counted at 885 regular intervals 886 -At study site only enough medication will be dispensed to reach next 887 appointment. All medication will be counted at visits and discussed at phone 888 encounters. 889 Procedure for return of used/unused trial products: 890 -Unused product will be properly destroyed at the site or returned to sponsor if 891 requested. 892 893 **Auxiliary Supply** 894 Subjects will use their own glucose monitors, lancet devices, and lancets. They will be 895 provided with log books. 896 Randomization 897 Treatment assignment will be made using stratified blocked randomization at visit 2. The 898 stratification variables will be prior insulin use and BMI (cut off 37 kg/m2). The 899 randomization code will be generated by the study statistician using SAS software, and 900 consecutively numbered envelopes will be created. The investigator opens the next 901 envelope at the randomization visit to determine the group assignment of the patient. 902 903 Blinding 904 This study is only blinded to the investigator performing the study assessments. The study is not blinded to the patient, nor the study doctor who will be providing diabetes

905 906 907

908

909

## **CONCOMITANT ILLNESSES AND MEDICATIONS:**

care to the patient and aid in insulin titration.

**Definitions:** 

- Oncomitant illness: any illness that is present at the start of the trial (i.e. at the first
- 911 *visit*).
- 912 Concomitant medication: any medication other than the trial product(s) that is taken
- 913 during the trial, including the screening and run-in periods.
- 914 Details of all concomitant illnesses and medication will be recorded at trial entry (i.e. at
- 915 the first visit). Any changes in concomitant medication will be recorded at each visit. If
- the change influences the subject's eligibility to continue in the trial, the Sponsor will be
- 917 informed.

- The information collected for each concomitant medication will include, at a minimum,
- 919 start date, stop date or continuing, and indication.
- 920 For each concomitant illness, date of onset, date of resolution or continuing, at a
- 921 minimum, will be recorded.

## **ADVERSE EVENTS AND PREGNANCY:**

- During each contact (phone or face-to-face) the subject will be asked about adverse
- events. All serious adverse events (SAE), suspected unexpected serious adverse
- 926 reactions (SUSAR), and serious adverse drug reactions (SADR) will be evaluated by the
- 927 investigator and recorded in the patients record. Other adverse events (AE) will be
- 928 evaluated and documented according to standard clinical practice
- The sponsor-investigator will collect the following information at minimum for each of
- 930 these events:
- 931 1. Study name
- 932 2. Patient identification (e.g. initials, sex, age)
- 933 3. Event (preferably a diagnosis)
- 934 4. Drug
- 935 5. Reporter identification (e.g. Name, or initials)
- 936 6. Causality
- 937 7. Outcome.

## 938 939

940

### **Definitions**

## 941 Adverse Event (AE):

- An AE is any undesirable medical event occurring to a subject in a clinical trial, whether or not related to the trial product(s). This includes events reported from the first trial
- related activity after the subject has signed the informed consent and until post treatment
- follow-up period as defined in the protocol. The following should not be recorded as
- 946 AEs, if recorded as medical history/concomitant illness on the CRF at screening:
- Pre-planned procedure, unless the condition for which the procedure was planned has worsened from the first trial related activity after the subject has signed the informed consent
  - Pre-existing conditions found as a result of screening procedures

## 951952

950

## **Clinical Laboratory Adverse Event:**

- A clinical laboratory AE is any clinical laboratory abnormality regarded as clinically
- 954 significant i.e. an abnormality that suggests a disease and/or organ toxicity and is of a

severity, which requires active management, (i.e. change of dose, discontinuation of trial product, more frequent follow-up or diagnostic investigation).

957 958

962

964

965

966

967

968

969

970

971

## **Serious Adverse Event (SAE):**

- A serious AE is an experience that at any dose results in any of the following:
- 960 Death
- A life-threatening\* experience
  - In-patient hospitalisation or prolongation of existing hospitalization
- A persistent or significant disability/incapacity
  - A congenital anomaly/birth defectSuspicion of transmission of infectious agents via the product.
  - Important medical events that may not result in death, be life-threatening\*, or require hospitalization may be considered an SAE when, based upon appropriate medical judgement, they may jeopardise the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition
  - \*The term life-threatening in the definition of SAE refers to an event in which the subject was at risk of death at the time of the event. It does not refer to an event which hypothetically might have caused death if it was more severe.

972973974

975

976

977

978

979

982

## **Serious Adverse Drug Reaction (SADR):**

An adverse drug reaction (ADR) is an adverse event for which a causal relationship (Possible/Probable relation) between the study drug and the occurrence of the event is suspected. The ADR should be classified as **serious** if it meets one or more of the seriousness criteria. Clinical judgement following thorough review of any event will be used to determine the relatedness of the event to the study drug.

980 981

#### **Non-Serious Adverse Event:**

A non-serious AE is any AE which does not fulfil the definition of an SAE.

983 984 985

986

987

#### **Severity Assessment Definitions:**

- Mild: Transient symptoms, no interference with the subject's daily activities
- Moderate: Marked symptoms, moderate interference with the subject's daily activities
- Severe: Considerable interference with the subject's daily activities, unacceptable

988 989 990

991

992

## **Relationship to study medication Assessment Definitions:**

- Probable: Good reasons and sufficient documentation to assume a causal relationship
- Possible: A causal relationship is conceivable and cannot be dismissed
  - Unlikely: The event is most likely related to an etiology other than the trial product

993994995

996

997

998

999

1000

#### **Outcome Categories and Definitions:**

- Recovered: Fully recovered or by medical or surgical treatment the condition has returned to the level observed at the first trial related activity after the subject signed the informed consent
- Recovering: The condition is improving and the subject is expected to recover from the event. This term should only be used when the subject has completed the trial

- Recovered with sequelae: As a result of the AE, the subject suffered persistent and significant disability/incapacity (e.g. became blind, deaf, paralysed). Any AE recovered with sequelae should be rated as an SAE
- 1004 Not recovered
- 1005 Fatal
- 1006 Unknown

## **Collection, Recording and Reporting of Adverse Events**

1009 All events meeting the definition of an adverse event will be collected and reported from 1010 the first trial related activity after the subject has signed the informed consent and until 1011 the end of the study. This will be monitored by an independent committee (see below). 1012 All serious and unexpected adverse events will be reported using FDA form 3500. All 1013 reports of SAEs/SAR/SUSARs or any events reported to the local health authorities must 1014 be sent to Novo Nordisk A/Swithin the same timeline used for reporting to regulatory 1015 authorities (see below). Further information about safety related events will be provided 1016 to Novo Nordisk A/S if specific requests are received.

1017 1018

1019 1020

1021

1022

1023

1024

1025

1026

1027

1028 1029

## **Data Safety Monitoring Board (DSMB)**

An independent DSMB will be set up for the trial to oversee safety and perform ongoing safety surveillance. The DSMB will be composed of 3 members who cover the relevant specialty as well as an independent statistician:

- Maria Ramos, MD (Endocrinology)
- Sumitha Hathiramani, MD (Endocrinology)
- Naim Maalouf, MD (Endocrinology)
- Song Zhang, PhD (Statistician)

The first meeting will occur after the enrolment of 15 subjects or three months after the first patient is enrolled, whichever comes first. The meetings will then occur on a quarterly basis, although the board may request more frequent meetings as needed. A formal report approved by all DSMB members will be sent to the PI and study coordinator within 3 weeks of the meeting and then forwarded to the IRB.

1030 1031 1032

1033

1034

1035

1036

1037

1038

All AEs will be presented at each meeting and will be available for informal review by the DSMB at any time after study initiation. All SAE and unanticipated but related AE will be promptly reported to the IRB (within 2 working days of PI's awareness for SAEs and within 10 working days for other reportable AEs). We intend to comply with all local legal, regulatory, and IRB requirements. We will also report to Novo Nordisk all SAEs, SUSARs, and SADRs at the same time such events are reported to regulatory authorities or within 15 working days from the sponsor-investigator becoming aware of such adverse events, whichever comes first.

1039 1040 1041

#### **Follow-up of Adverse Events**

During and following a subject's participation in a clinical trial, the sponsor-investigator and institution will provide adequate medical care to the study subject for any study-related adverse events, including clinically significant laboratory values related to the study. This medical care for study subjects will be provided regardless of their insurance status.

- All adverse events classified as serious or severe or possibly/probably related to the trial
- product must be followed until the subject has recovered and all queries have been
- resolved. For cases of chronic conditions follow-up until the outcome category is
- "recovered" is not required, as these cases can be closed with an outcome of "recovering"
- or "not recovered".
- All other adverse events must be followed until the outcome of the event is "recovering"
- 1053 (for chronic conditions), or "recovered" or until the end of study, whichever comes first,
- and until all queries related to these AEs have been resolved.

## 1056 Pregnancy

- Study subjects will be instructed to notify the sponsor-investigator immediately if they
- become pregnant. If using liraglutide this medication will be discontinued immediately.

1059 1060

1061

The sponsor-investigator will report to Novo Nordisk any pregnancy occurring during the trial period. Reporting of pregnancy by sponsor-investigator should occur within the same timelines described above for reporting of Adverse Events.

1062 1063 1064

1065

Pregnancy complications will be recorded as adverse event(s). If the infant has a congenital anomaly/birth defect this must be reported and followed up as a serious adverse event.

1066 1067 1068

1069

1070

1071

### Precautions/Over-dosage

- The following precautions and procedures will be observed in the event of overdose by any trial product provided during the study: if asymptomatic, the patient is instructed to call the study doctor immediately after discovering the overdosage and obtain case-specific instructions; if symptomatic, the patient is instructed to call the EMS for
- specific instructions; if symptomatic, the patient is instructed to call the EMS function immediate treatment.

1074

10/4

1076

1077

1078

1079

## **LIABILITY AND SUBJECT INSURANCE:**

During and following a subject's participation in trial, the sponsor-investigator and his/her institution will provide adequate medical care to the study subject for any study-related adverse events, including clinically significant laboratory values related to the study. This medical care for study subjects will be provided regardless of their insurance status.

- The sponsor-investigator will be responsible for the conduct of the study and that the sponsor-investigator agrees to defend, indemnify, and hold harmless Novo Nordisk, as
- sponsor-investigator agrees to defend, indemnify, and hold harmless Novo Nordisk, any of its parent companies, affiliates, or subsidiaries, and their respective officers, directors,
- 1085 employees, agents, representatives, distributors, salespersons, customers, licensees, and
- end-users from and against any claim, suit, demand, loss, damage, expense or liability
- imposed by any third party arising from or related to: (a) any breach of sponsor-
- investigator's obligations; or (b) sponsor-investigator's negligent or grossly negligent use
- or willful misuse of the study drug, the results, or services derived therefrom. This
- indemnification shall not apply in the event and to the extent that a court of competent
- jurisdiction or a duly appointed arbiter determines that such losses or liability arose as a

result of Novo Nordisk's gross negligence, intentional misconduct, or material breach of its responsibilities.

1094 1095

1097

1098

## **EVALUABILITY OF SUBJECTS:**

All patients and collected data will be included in the intention to treat analysis.

A secondary confirmatory analysis will be performed using only completers data, where all data from patients with an overall compliance rate during the study period of <50%

will be excluded. The subjects and observations to be excluded, and the reasons for their exclusion will be documented and signed by those responsible prior to database release.

The documentation must be stored together with the remaining trial documentation.

1101 1102 1103

## PREMATURE TERMINATION OF STUDY:

Study can be discontinued if funding is withdrawn or by the Data Safety Monitoring

Board (DSMB) if there is evidence of futility or excess harm. The study statistician will

monitor the data quarterly and discuss any observed trends with the other members of the

DSMB who will make such decision following pre-established guidelines.

1107 1108 1109

## **PUBLICATION PLAN:**

- We plan to publish the data from this clinical trial in peer reviewed scientific journals
- 1111 (i.e. Diabetes Care). We anticipate at least two manuscripts to results from this work
- 1112 (possibly one on clinical efficacy and safety, one on healthcare utilization and cost
- data). We expect the final manuscripts to be completed around December 1<sup>st</sup>, 2016. All
- manuscripts will be submitted to Novo Nordisk for review and commenting 1 month
- before external submission. We also plan to present the data at the American Diabetes
- 1116 Association and/or The Endocrine Society scientific meetings as poster or oral
- 1117 presentations.
- We have registered the study with clinicaltrials.gov.

#### **REFERENCES:**

- 1. CDC. *National Diabetes Fact Sheet 2011*. 2013 [cited 2013 07/05/2013]; Available from: http://www.cdc.gov/diabetes/pubs/pdf/ndfs 2011.pdf.
- Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet, 1998. 1127 352(9131): p. 837-53.
- Holman, R.R., et al., 10-year follow-up of intensive glucose control in type 2 diabetes. N Engl J Med, 2008. **359**(15): p. 1577-89.
- Ohkubo, Y., et al., Intensive insulin therapy prevents the progression of diabetic microvascular complications in Japanese patients with non-insulin-dependent diabetes mellitus: a randomized prospective 6-year study. Diabetes Res Clin Pract, 1995. 28(2): p. 103-17.
- Shichiri, M., et al., Long-term results of the Kumamoto Study on optimal diabetes control in type 2 diabetic patients. Diabetes Care, 2000. 23 Suppl 2: p. B21-9.
- 1136 6. Stark Casagrande, S., et al., *The Prevalence of Meeting A1C, Blood Pressure, and LDL Goals Among People With Diabetes, 1988-2010.* Diabetes Care, 2013.
- 1138 7. McWilliams, J.M., et al., Differences in control of cardiovascular disease and diabetes by race, ethnicity, and education: U.S. trends from 1999 to 2006 and effects of medicare coverage. Ann Intern Med, 2009. **150**(8): p. 505-15.
- Saydah, S.H., J. Fradkin, and C.C. Cowie, *Poor control of risk factors for* vascular disease among adults with previously diagnosed diabetes. JAMA, 2004. **291**(3): p. 335-42.
- American Diabetes, A., *Economic costs of diabetes in the U.S. In 2007.* Diabetes Care, 2008. **31**(3): p. 596-615.
- Herman, W.H., *The economic costs of diabetes: is it time for a new treatment paradigm?* Diabetes Care, 2013. **36**(4): p. 775-6.
- 1148 11. Li, R., et al., Medical costs associated with type 2 diabetes complications and comorbidities. Am J Manag Care, 2013. **19**(5): p. 421-30.
- 1150 12. Inzucchi, S.E., et al., Management of hyperglycaemia in type 2 diabetes: a
  1151 patient-centered approach. Position statement of the American Diabetes
  1152 Association (ADA) and the European Association for the Study of Diabetes
  1153 (EASD). Diabetologia, 2012. **55**(6): p. 1577-1596.
- 13. Garber, A.J., *Methods to enhance delivery of prandial insulin and basal-prandial insulin.* Diabetes Obes Metab, 2013. **15 Suppl 1**: p. 11-7.
- 1156 14. Lamanna, C., et al., Effect of metformin on cardiovascular events and mortality: a
  1157 meta-analysis of randomized clinical trials. Diabetes Obes Metab, 2011. **13**(3): p.
  1158 221-8.
- 1159 15. Simonson GD, C.R., Reader D, Bergenstal RM, International Diabetes Center treatment of type 2 diabetes glucose
- 1161 *algorithm*. Diabetes Management, 2011. 1: p. 175–189.
- 1162 16. Bergenstal, R.M., et al., Adjust to target in type 2 diabetes: comparison of a simple algorithm with carbohydrate counting for adjustment of mealtime insulin glulisine. Diabetes Care, 2008. **31**(7): p. 1305-10.

- 1165 17. Blonde, L., et al., Patient-directed titration for achieving glycaemic goals using a
  1166 once-daily basal insulin analogue: an assessment of two different fasting plasma
  1167 glucose targets the TITRATE study. Diabetes Obes Metab, 2009. 11(6): p. 6231168 31.
- 1169 18. Davidson, M.B., et al., A stepwise approach to insulin therapy in patients with type 2 diabetes mellitus and basal insulin treatment failure. Endocr Pract, 2011. 17(3): p. 395-403.
- 1172 19. Garber, A.J., *Treat-to-target trials: uses, interpretation and review of concepts.*1173 Diabetes Obes Metab, 2013.
- Hermansen, K., et al., A 26-week, randomized, parallel, treat-to-target trial comparing insulin detemir with NPH insulin as add-on therapy to oral glucose-lowering drugs in insulin-naive people with type 2 diabetes. Diabetes Care, 2006. 29(6): p. 1269-74.
- Holman, R.R., et al., *Three-year efficacy of complex insulin regimens in type 2 diabetes.* N Engl J Med, 2009. **361**(18): p. 1736-47.
- Jabbour, S., *Primary care physicians and insulin initiation: multiple barriers, lack of knowledge or both?* Int J Clin Pract, 2008. **62**(6): p. 845-7.
- Lankisch, M.R., et al., Introducing a simplified approach to insulin therapy in type 2 diabetes: a comparison of two single-dose regimens of insulin glulisine plus insulin glargine and oral antidiabetic drugs. Diabetes Obes Metab, 2008. 10(12): p. 1178-85.
- Meneghini, L., et al., Comparison of 2 intensification regimens with rapid-acting insulin aspart in type 2 diabetes mellitus inadequately controlled by once-daily insulin detemir and oral antidiabetes drugs: the step-wise randomized study.

  Endocr Pract, 2011. 17(5): p. 727-36.
- Rosenstock, J., et al., Advancing insulin therapy in type 2 diabetes previously treated with glargine plus oral agents: prandial premixed (insulin lispro protamine suspension/lispro) versus basal/bolus (glargine/lispro) therapy.

  Diabetes Care, 2008. **31**(1): p. 20-5.
- 1194 26. Umpierrez, G.E., et al., Randomized Study Comparing a Basal Bolus With a Basal 1195 Plus Correction Insulin Regimen for the Hospital Management of Medical and 1196 Surgical patients With Type 2 Diabetes: Basal Plus Trial. Diabetes Care, 2013.
- 1197 27. Rossetti, L., et al., Effect of chronic hyperglycemia on in vivo insulin secretion in partially pancreatectomized rats. J Clin Invest, 1987. **80**(4): p. 1037-44.
- Del Prato, S., Role of glucotoxicity and lipotoxicity in the pathophysiology of Type 2 diabetes mellitus and emerging treatment strategies. Diabet Med, 2009. **26**(12): p. 1185-92.
- 1202 29. Henry, R.R., et al., *Intensive conventional insulin therapy for type II diabetes*.

  1203 *Metabolic effects during a 6-mo outpatient trial*. Diabetes Care, 1993. **16**(1): p.
  1204 21-31.
- 1205 30. Intensive Blood Glucose Control and Vascular Outcomes in Patients with Type 2
  1206 Diabetes. New England Journal of Medicine, 2008. **358**(24): p. 2560-2572.
- 1207 31. Charbonnel, B., et al., *Insulin therapy for diabetes mellitus: treatment regimens* and associated costs. Diabetes Metab, 2012. **38**(2): p. 156-63.
- 1209 32. Effects of Intensive Glucose Lowering in Type 2 Diabetes. New England Journal of Medicine, 2008. **358**(24): p. 2545-2559.

- 1211 33. Pi-Sunyer, F.X., Weight loss and mortality in type 2 diabetes. Diabetes Care, 2000. **23**(10): p. 1451-2.
- Williamson, D.F., et al., *Intentional weight loss and mortality among overweight individuals with diabetes.* Diabetes Care, 2000. **23**(10): p. 1499-504.
- 1215 35. Defronzo, R.A., Banting Lecture. From the triumvirate to the ominous octet: a
  1216 new paradigm for the treatment of type 2 diabetes mellitus. Diabetes, 2009. **58**(4):
  1217 p. 773-95.
- J., B., et al. Weight gain within the first year after new onset diabetes is
   associated with risk of cardiovascular mortality: A cohort of 8326 primary care
   patients. in European Association for the Study of Diabetes 2012 Meeting. 2012.
   Berlin, Germany.
- 1222 37. Anderson, R.T., et al., *Effect of intensive glycemic lowering on health-related*1223 quality of life in type 2 diabetes: ACCORD trial. Diabetes Care, 2011. **34**(4): p.
  1224 807-12.
- 1225 38. Giordano, C., *Insulin therapy: unmet needs and new perspectives.* Minerva Endocrinol, 2013. **38**(1): p. 95-102.
- 1227 39. Henry, R.R., et al., Efficacy of antihyperglycemic therapies and the influence of baseline hemoglobin A(1C): a meta-analysis of the liraglutide development program. Endocr Pract, 2011. 17(6): p. 906-13.
- 40. Avramidis, I., et al., Optimizing Glycemic Control in T2DM Patients Previously
   Treated with Intensive Insulin Therapy and Switched to Exenatide-Insulin
   Glargine Combination. Diabetes, 2013. 62(Supplement 1): p. A217-A364.
- 41. Blase, E.B., S; Li, Y; Grimm, M, Add-On Treatment with Exenatide Once Weekly
  vs. Daily Basal Insulin in Patients with A1C ≥8.5%. Diabetes, 2013.
  62(Supplement 1): p. A217-A364.
- Trautmann, M.V.g., L., Guerci, B.; Stranks, S.; Han, J.; Malloy, J.; Boadman, M.;
   Diaman, M., Exenatide Once Weekly: Sustained Glycemic and Weight Control
   Through 3 Years Compared with Insulin Glargine. Diabetes, 2013.
   62(Supplement 1): p. A1-A98.
- 1240 43. Riddle, M.S., Y, Cariou, B.; Huelgas, R.G.; Roy-Duval, C; Hecquet, C.; Digenio, A.; Rosenstock, J, Once-daily lixisenatide as add-on to basal insulin ± OADs in patients with Type 2 diabetes selectively reduces postprandial hyperglycemic daytime exposure. Diabetes, 2013. **62**(Supplement 1): p. A217-A364.
- 1244 44. Rosenstock, J., et al., Expanding the Basal-Plus Regimen: Basal Insulin +
  1245 Lixisenatide is More Likely to Achieve the Composite Outcome of Hba1c<7%, No
  1246 Documented Symptomatic Hypoglycemia and No Weight Gain Compared with
  1247 Basal + Prandial Insulin. Diabetes, 2013. 62(Supplement 1): p. A217-A364.
- 1248 45. Diamant, M.N., M.; Shaginian, R.; Malone, J.; Cleall, S.; De Vries, D.; Hoogwerf, B; Macconell, L; Wolffenbuttel, B., Exenatide BID vs. Insulin Lispro TIDM
  1250 Added to Titrated Insulin Glargine QD in Metformin-Treated T2DM Patients
  1251 Resulted in Similar Glycemic Control but Weight Loss and Less Hypoglycemia:
- 1252 The 4B Study. Diabetes, 2013. 62(Supplement 1): p. A1-A98.
  1253 46. Balena, R., et al., Combination therapy with GLP-1 receptor agonists and basal insulin: a systematic review of the literature. Diabetes, Obesity and Metabolism,

1255 2013. **15**(6): p. 485-502.

- Mathiel, C.R., H; Cariou, B, Handelsman, Y; Philis-Tsimikas, A; Francisco, A;
   Rana, A; Zinman, B, Comparison of Addition of Liraglutide to Insulin Degludec
   Plus Metformin vs. Addition of a Single Dose of Rapid-Acting Insulin Analog to
   Largest Meal in Type-2 Diabetes. Diabetes, 2013. 62(Supplement 1): p. A217 A364.
- 1261 48. DeVries, J.H., et al., Sequential intensification of metformin treatment in type 2 1262 diabetes with liraglutide followed by randomized addition of basal insulin 1263 prompted by A1C targets. Diabetes Care, 2012. **35**(7): p. 1446-54.
- 1264 49. Macconell, L., et al., *Exenatide once weekly: sustained improvement in glycemic control and cardiometabolic measures through 3 years*. Diabetes Metab Syndr Obes, 2013. **6**: p. 31-41.
- 1267 50. Chaudhary, M.A. and S.C. Stearns, *Estimating confidence intervals for cost-*1268 effectiveness ratios: an example from a randomized trial. Stat Med, 1996. **15**(13):
  1269 p. 1447-58.